CLINICAL TRIAL: NCT00167830
Title: Understanding The Barriers in Treatment of Obesity in Adolescents 11-18 in Central Virginia
Brief Title: Barriers to Treatment in Obese Adolescents
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: VA Premier Health (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 760
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Obesity
Keywords: Pediatric Overweight,; African American;; Adolescent;; Intervention,; Teasing;; Self-esteem; Quality of Life; Metabolic syndrome; Insulin resistance; Diabetes; Nutrition; Motivation; Culture; BMI; Cardiorespiratory fitness; Resistance Training; Compliance
MeSH Terms: conditions — Obesity; Metabolic Syndrome; Insulin Resistance; Diabetes Mellitus; Patient Compliance | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lifestyle Intervention (Experimental): Dietary modification and exercise.
  Interventions: Behavioral: Motivational Interviewing; Behavioral: Strength and Cardiovascular Conditioning; Behavioral: Food selection and portion control

INTERVENTIONS:
Behavioral: Motivational Interviewing — Biweekly meetings with a behavior specialist to review subject's progress with the protocol and explore challenges subject is facing in adopting healthy lifestyle behaviors.
Behavioral: Strength and Cardiovascular Conditioning — Subjects take part in an exercise program to include 30 minutes of cardiorespiratory exercise at 70% maximum heart rate, and 30 minutes of strength training on Nautilus machines.
Behavioral: Food selection and portion control — Subjects meet on a biweekly basis with a registered dietitian who presents educational information about healthy food selection and portion control.

SUMMARY:
The purpose of this study is to identify significant racial and ethnical differences in risk factors for development of obesity and weight loss in adolescents in Central Virginia

DETAILED DESCRIPTION:
* Participation for 6 months in a program incorporating exercise, nutritional counseling and behavioral support leads to measurable improvements in overall fitness, metabolic indicators and loss of body fat for obese adolescents.
* Degree of loss of body fat, improved overall fitness and improvements in metabolic indicators can be correlated with the degree of compliance and participation for 6 months in the program.
* Parental involvement and support can be correlated with the degree of compliance and participation in the program.
* Socioeconomic factors can be correlated with the degree of compliance and participation in the program.
* Cultural differences in diet, attitudes toward body shape, and family dynamics can be correlated with success or failure in a weight loss program.
* Individual differences in self-esteem, self-discipline and feelings of connectedness with family members can be correlated with success or failure in a weight loss program.

ELIGIBILITY:
Inclusion Criteria:

* Age 11-18
* Above 95th percentile for weight
* Reside within 30 miles of program site
* Ability to comprehend basic instructions
* Ability to perform basic exercise movements

Exclusion Criteria:

* Having a metabolic disorder that causes weight gain
* Having a cognitive deficit that impacts learning and comprehension
* Having a physical defect that prevents exercise

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 292 (Actual)
Dates: Start 2003-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
A decrease in body mass index. | 6 months and 1 year
Improvement in metabolic indicators. | 6 months and 1 year
Improvement in fitness measures | 6 months and 1 year

SECONDARY OUTCOMES:
Improved subject compliance with exercise and diet. | 6 months and 1 year
Improved parental compliance and support. | 6 months and 1 year
Increase knowledge of nutritional principles | 6 months and 1 year
Improved attitude toward healthy behaviors | 6 months and 1 year
Increased self-esteem and motivation | 6 months and 1 year
Decreased negativity | 6 months and 1 year
Improved family cohesiveness | 6 months and 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Edmond Wickham, M.D., Principal Investigator — Virginia Commonwealth University Depts. of Internal Medicine and Pediatrics
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- [Background] Wickham EP, Stern M, Evans RK, Bryan DL, Moskowitz WB, Clore JN, Laver JH. Prevalence of the metabolic syndrome among obese adolescents enrolled in a multidisciplinary weight management program: clinical correlates and response to treatment. Metab Syndr Relat Disord. 2009 Jun;7(3):179-86. doi: 10.1089/met.2008.0038. PMID 19450141
- [Background] Porter JS, Bean MK, Gerke CK, Stern M. Psychosocial factors and perspectives on weight gain and barriers to weight loss among adolescents enrolled in obesity treatment. J Clin Psychol Med Settings. 2010 Jun;17(2):98-102. doi: 10.1007/s10880-010-9186-3. PMID 20119710
- [Background] Bean MK, Mazzeo SE, Stern M, Evans RK, Bryan D, Ning Y, Wickham EP 3rd, Laver J. Six-month dietary changes in ethnically diverse, obese adolescents participating in a multidisciplinary weight management program. Clin Pediatr (Phila). 2011 May;50(5):408-16. doi: 10.1177/0009922810393497. Epub 2011 Jan 10. PMID 21224253
- [Result] Stern M, Mazzeo SE, Gerke CK, Porter JS, Bean MK, Laver JH. Gender, ethnicity, psychosocial factors, and quality of life among severely overweight, treatment-seeking adolescents. J Pediatr Psychol. 2007 Jan-Feb;32(1):90-4. doi: 10.1093/jpepsy/jsl013. Epub 2006 Jul 3. PMID 16818482
- [Result] Stern M, Mazzeo SE, Porter J, Gerke C, Bryan D,and Laver J. Self-esteem, teasing and quality of life: African American adolescent girls participating in a family-based pediatric overweight intervention. Journal of Clinical Psychology in Medical Settings. DOI:10.1007/s10880-006-9029-4, 2006
- [Derived] Browning MG, Bean MK, Wickham EP, Stern M, Evans RK. Cardiometabolic and Fitness Improvements in Obese Girls Who Either Gained or Lost Weight during Treatment. J Pediatr. 2015 Jun;166(6):1364-9. doi: 10.1016/j.jpeds.2015.03.011. Epub 2015 Apr 15. PMID 25890676
- [Derived] Ning Y, Yang S, Evans RK, Stern M, Sun S, Francis GL, Wickham EP 3rd. Changes in body anthropometry and composition in obese adolescents in a lifestyle intervention program. Eur J Nutr. 2014 Jun;53(4):1093-102. doi: 10.1007/s00394-013-0612-9. Epub 2013 Nov 10. PMID 24212451